CLINICAL TRIAL: NCT01610752
Title: Expecting Success: Personalized Management of Body Weight During Pregnancy
Brief Title: Personalized Management of Body Weight During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Leanne Redman, Principal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PBRC 11024; U01DK094418-01 (NIH)
Record Dates: First submitted 2012-05-31; First posted 2012-06-04 (Estimated); Results first posted 2018-12-12 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-08

CONDITIONS: Weight Gain During Pregnancy
Keywords: Pregnancy; Gestational weight gain
MeSH Terms: conditions — Gestational Weight Gain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- SmartMoms-Clinic (Experimental): If picked for this group, you will attend study meetings with a weight management counselor. During the second trimester study meetings occur 4 times per month. During the third trimester you will attend study meetings 2 times per month. These meetings will cover many topics to help you learn about weight management during pregnancy. You will be taught how to use different tools provided to help you monitor your weight. We will ask you to record your body weight (using a scale we will provide) as well as your food intake and exercise habits.
  Interventions: Behavioral: SmartMoms
- SmartMoms-Phone (Experimental): If picked for this group, you will have two individual sessions with a weight management counselor. At the first session, you will receive a scale and other technology to help manage your weight during pregnancy. Each week you will receive information from a weight management counselor via a Smartphone (you can use your own Smartphone or one will be provided to you). The information will cover topics to help manage your weight during pregnancy. You will be taught how to use different tools provided to help you monitor your weight. We will ask you to measure your body weight (using a scale we will provide) as well as monitor your food intake and exercise habits with the Smartphone.
  Interventions: Behavioral: SmartMoms
- Physician Directed (No Intervention): If picked for this group, you will receive weight management advice from your physician's office.

INTERVENTIONS:
Behavioral: SmartMoms — This intervention will cover many topics to help you learn about weight management during pregnancy. You will be taught how to use different tools provided to help you monitor your weight. We will ask you to record your body weight (using a scale we will provide) as well as your food intake and exercise habits.
  Arms: SmartMoms-Clinic; SmartMoms-Phone

SUMMARY:
The purpose of this study is to determine how to help manage weight gain during pregnancy. This study is part of the National Consortium 'LIFE-Moms: Lifestyle interventions in expectant moms'. LIFE-Moms is 7 studies funded to test different lifestyle interventions in overweight and obese pregnant women.

DETAILED DESCRIPTION:
The study will last 22 months, from screening until study completion. The entire study will include 3 screening visits, receipt of weight management advice, second trimester testing, third trimester testing and three follow up visits during the first year after the baby is born. Participants will randomly be assigned to 1 of 3 programs to help manage their weight during pregnancy:

1. Physician Directed group
2. SmartMoms-Clinic group
3. SmartMoms-Phone group

ELIGIBILITY:
Inclusion Criteria:

* Are pregnant.
* Are between 18 and 40 years old.
* Have a BMI (a number calculated from your height and weight) equal to or above 25kg/m2.
* Establish prenatal care before 12 weeks of your pregnancy.
* Can read, speak and understand English.

Exclusion Criteria:

* Do not plan to deliver your baby at Woman's Hospital, Baton Rouge, LA
* Are pregnant with more than one infant.
* Have habitually smoked during the last 6 months.
* Currently abuse or have abused illegal or prescription drugs in the last 6 months.
* Consume more than 2 alcoholic drinks per week.
* Are unwilling to avoid pregnancy for 12 months following delivery.
* Are unwilling to enroll your baby in the 12 month follow-up testing planned in this study.
* Are planning to move out of the area within the next 2 years or plan to be out of the study area for more than 1 month in the next year.
* Are unwilling to be assigned at random to any of the intervention groups.
* Are planning to terminate your pregnancy.
* Are planning to give your baby up for adoption.
* Are pregnant with a baby who has a known fetal anomaly.
* Have a reason that exercising is unsafe (determined by your physician or study staff).
* Have had or plan to have bariatric surgery within 1 year of your expected delivery.
* Currently have or have a history of the following:
* 3 or more first trimester miscarriages
* High blood pressure
* Type 1 diabetes
* Diagnosis of pregnancy related diabetes during screening
* HIV or AIDS
* Psychotic disorder, major depressive episode, bipolar disorder or eating disorder
* Any other pregnancy, blood, heart, lung, hormone, or digestive problem that your doctor considers unsafe for participation in this study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leanne M Redman, Ph.D., Principal Investigator — Pennington Biomedical Research Center
Locations (2):
- United States (2):
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Woman's Hospital, Baton Rouge, Louisiana

REFERENCES:
- [Derived] Cabre HE, Drews KL, Pomeroy J, Keadle SK, Arteaga SS, Franks PW, Haire-Joshu D, Knowler WC, Pi-Sunyer X, Van Horn L, Wing RR, Cahill AG, Clifton RG, Couch KA, Gallager D, Josefson JL, Joshipura K, Klein S, Martin CK, Peaceman AM, Phelan S, Thom EA, Redman LM; LIFE-Moms Research Group. LIFE-Moms: effects of multicomponent lifestyle randomized control trial on physical activity during pregnancy in women with overweight and obesity. Int J Behav Nutr Phys Act. 2025 Sep 30;22(1):119. doi: 10.1186/s12966-025-01805-9. PMID 41029405
- [Derived] Flanagan EW, Drews KL, Cade WT, Franks PW, Gallagher D, Phelan S, Van Horn L, Redman LM. Metabolic Health and Heterogenous Outcomes of Prenatal Interventions: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2025 Aug 1;8(8):e2528264. doi: 10.1001/jamanetworkopen.2025.28264. PMID 40839263
- [Derived] Redman LM, Drews KL, Klein S, Horn LV, Wing RR, Pi-Sunyer X, Evans M, Joshipura K, Arteaga SS, Cahill AG, Clifton RG, Couch KA, Franks PW, Gallagher D, Haire-Joshu D, Martin CK, Peaceman AM, Phelan S, Thom EA, Yanovski SZ, Knowler WC; LIFE-Moms Research Group. Attenuated early pregnancy weight gain by prenatal lifestyle interventions does not prevent gestational diabetes in the LIFE-Moms consortium. Diabetes Res Clin Pract. 2021 Jan;171:108549. doi: 10.1016/j.diabres.2020.108549. Epub 2020 Nov 22. PMID 33238176
- [Derived] Palmer MJ, Henschke N, Bergman H, Villanueva G, Maayan N, Tamrat T, Mehl GL, Glenton C, Lewin S, Fonhus MS, Free C. Targeted client communication via mobile devices for improving maternal, neonatal, and child health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013679. doi: 10.1002/14651858.CD013679. PMID 32813276
- [Derived] Altazan AD, Redman LM, Burton JH, Beyl RA, Cain LE, Sutton EF, Martin CK. Mood and quality of life changes in pregnancy and postpartum and the effect of a behavioral intervention targeting excess gestational weight gain in women with overweight and obesity: a parallel-arm randomized controlled pilot trial. BMC Pregnancy Childbirth. 2019 Jan 29;19(1):50. doi: 10.1186/s12884-019-2196-8. PMID 30696408
- [Derived] Peaceman AM, Clifton RG, Phelan S, Gallagher D, Evans M, Redman LM, Knowler WC, Joshipura K, Haire-Joshu D, Yanovski SZ, Couch KA, Drews KL, Franks PW, Klein S, Martin CK, Pi-Sunyer X, Thom EA, Van Horn L, Wing RR, Cahill AG; LIFE-Moms Research Group. Lifestyle Interventions Limit Gestational Weight Gain in Women with Overweight or Obesity: LIFE-Moms Prospective Meta-Analysis. Obesity (Silver Spring). 2018 Sep;26(9):1396-1404. doi: 10.1002/oby.22250. Epub 2018 Sep 6. PMID 30230252
- [Derived] Redman LM, Gilmore LA, Breaux J, Thomas DM, Elkind-Hirsch K, Stewart T, Hsia DS, Burton J, Apolzan JW, Cain LE, Altazan AD, Ragusa S, Brady H, Davis A, Tilford JM, Sutton EF, Martin CK. Effectiveness of SmartMoms, a Novel eHealth Intervention for Management of Gestational Weight Gain: Randomized Controlled Pilot Trial. JMIR Mhealth Uhealth. 2017 Sep 13;5(9):e133. doi: 10.2196/mhealth.8228. PMID 28903892
- [Derived] Sutton EF, Cain LE, Vallo PM, Redman LM. Strategies for Successful Recruitment of Pregnant Patients Into Clinical Trials. Obstet Gynecol. 2017 Mar;129(3):554-559. doi: 10.1097/AOG.0000000000001900. PMID 28178062
- [Derived] Clifton RG, Evans M, Cahill AG, Franks PW, Gallagher D, Phelan S, Pomeroy J, Redman LM, Van Horn L; LIFE-Moms Research Group. Design of lifestyle intervention trials to prevent excessive gestational weight gain in women with overweight or obesity. Obesity (Silver Spring). 2016 Feb;24(2):305-13. doi: 10.1002/oby.21330. Epub 2015 Dec 26. PMID 26708836

RESULTS

PARTICIPANT FLOW:
Groups:
- SmartMoms-Phone: If picked for this group, you will have two individual sessions with a weight management counselor. At the first session, you will receive a scale and other technology to help manage your weight during pregnancy. Each week you will receive information from a weight management counselor via a Smartphone (you can use your own Smartphone or one will be provided to you). The information will cover topics to help manage your weight during pregnancy. We will ask you to measure your body weight (using a scale we will provide) as well as monitor your food intake and exercise habits with the Smartphone.
  SmartMoms: This intervention will cover many topics to help you learn about weight management during pregnancy. You will be taught how to use different tools provided to help you monitor your weight. We will ask you to record your body weight (using a scale we will provide) as well as your food intake and exercise habits.
Period: Overall Study
Arm/Group | SmartMoms-Clinic | SmartMoms-Phone | Physician Directed
Started | 18 | 19 | 17
Completed | 18 | 19 | 13
Not Completed | 0 | 0 | 4
Not completed — Miscarriage/Pregnancy loss | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SmartMoms-Clinic | SmartMoms-Phone | Physician Directed | Total
Number analyzed (Participants) | 18 | 19 | 17 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.2 (4.8) | 29.0 (4.2) | 29.5 (5.1) | 29.2 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 17 | 54
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 2 | 6 | 13
  White | 11 | 16 | 11 | 38
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Parity [Mean (Standard Deviation); unit: viable pregnancies] — Parity is the number of pregnancies that have reached viability. Appropriate individual scores are 0, 1, 2, etc. Means and standard deviations include decimal numbers.
  viable pregnancies | 0.7 (0.8) | 0.9 (1.1) | 0.6 (0.5) | 0.8 (0.8)
Pregravid BMI [Count of Participants; unit: Participants]
  Overweight (25.0-29.9 kg/m2) | 8 | 8 | 9 | 25
  Obese (30.0-40.0 kg/m2) | 10 | 11 | 8 | 29
Family income per year [Count of Participants; unit: Participants]
  <$5000-$39,999 | 9 | 7 | 7 | 23
  $40,000-$99,999 | 7 | 5 | 5 | 17
  ≥$100,000 | 2 | 7 | 5 | 14
Education [Count of Participants; unit: Participants]
  Some high school | 1 | 0 | 0 | 1
  High school diploma/GED/1-3 years of college | 5 | 6 | 7 | 18
  College degree | 7 | 11 | 4 | 22
  Postgraduate work | 5 | 2 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Count of Women Who Have Excess Gestational Weight Gain
Description: Count of pregnant women who gain more weight during pregnancy than is recommended by the Institute of Medicine Gestational Weight Gain guidelines
Time Frame: Approximately 6 months (from 10-13 weeks gestation to 35-36 weeks gestation)
Measure: Count of Participants; unit: Participants
Arm/Group | SmartMoms-Clinic | SmartMoms-Phone | Physician Directed
Number analyzed (Participants) | 18 | 19 | 13
Participants | 10 | 11 | 11

2. Secondary Outcome: Total Gestational Weight Gain
Time Frame: Approximately 6 months (from 10-13 weeks gestation to 35-36 weeks gestation)
Measure: Least Squares Mean (Standard Error); unit: kilograms
Arm/Group | SmartMoms-Clinic | SmartMoms-Phone | Physician Directed
Number analyzed (Participants) | 18 | 19 | 13
kilograms | 8.0 (1.3) | 10.0 (1.2) | 12.8 (1.5)

3. Secondary Outcome: Gestational Weight Gain Per Week
Description: "per week" is included to adjust for the different length of time between weight measurements
Time Frame: Approximately 6 months (from 10-13 weeks gestation to 35-36 weeks gestation)
Measure: Least Squares Mean (Standard Error); unit: kilograms per week
Arm/Group | SmartMoms-Clinic | SmartMoms-Phone | Physician Directed
Number analyzed (Participants) | 18 | 19 | 13
kilograms per week | 0.31 (0.05) | 0.39 (0.05) | 0.49 (0.06)

4. Post Hoc Outcome: Intervention Cost for Participant
Description: Costs incurred for travel to and from treatment sessions and time spent with the counselor while accounting for session attendance and intervention adherence. Outcome measure only assessed in SmartMoms-Clinic and SmartMoms-Phone groups because the Physician Directed group did not receive any intervention.
Time Frame: Approximately 6 months (from 1st trimester until delivery)
Measure: Mean (Standard Deviation); unit: US dollars
Arm/Group | SmartMoms-Clinic | SmartMoms-Phone
Number analyzed (Participants) | 18 | 19
US dollars | 347 (40) | 97 (6)

5. Post Hoc Outcome: Percentage of Days With Intervention Adherence
Description: Adherence to the SmartMoms intervention was defined as the percentage of days participants weighed and recorded step counts in comparison to the expected number of days. Outcome measure only assessed in SmartMoms-Clinic and SmartMoms-Phone groups because the Physician Directed group did not receive any intervention.
Time Frame: Approximately 6 months (from 1st trimester until delivery)
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | SmartMoms-Clinic | SmartMoms-Phone
Number analyzed (Participants) | 18 | 19
percentage of days | 60.8 (6.4) | 76.5 (4.5)

6. Post Hoc Outcome: Intervention Cost for Clinic
Description: Clinic costs included interventionist time for training, session preparation, participant contacts, routine staff meetings, and scale and pedometer cost. Outcome measure only assessed in SmartMoms-Clinic and SmartMoms-Phone groups because the Physician Directed group did not receive any intervention. The US dollar cost was standard across each participant in each group so there is $0 standard deviation.
Time Frame: Approximately 6 months (from 1st trimester until delivery)
Measure: Mean (Standard Deviation); unit: US dollars
Arm/Group | SmartMoms-Clinic | SmartMoms-Phone
Number analyzed (Participants) | 18 | 19
US dollars | 419 (0.0) | 215 (0.0)

ADVERSE EVENTS:
Time Frame: Approximately 6 months (10-13 weeks gestation to delivery)
Arm/Group | SmartMoms-Clinic | SmartMoms-Phone | Physician Directed
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/19 | 0/17
Serious Adverse Events (participants affected / at risk) | 2/18 | 1/19 | 5/17
Other Adverse Events (participants affected / at risk) | 13/18 | 15/19 | 12/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SmartMoms-Clinic (N=18) | SmartMoms-Phone (N=19) | Physician Directed (N=17)
Miscarriage/pregnancy loss (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 4 (4)
Kidney stones requiring hospitalization (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration due to Crohn's disease requiring hospitalization (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia requiring hospitalization (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Severe pre-eclampsia requiring hospitalization (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SmartMoms-Clinic (N=18) | SmartMoms-Phone (N=19) | Physician Directed (N=17)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (3)
Anemia (Blood and lymphatic system disorders) | 3 (3) | 4 (4) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 6 (7) | 2 (3)
Cold/sinus congestion (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 3 (3) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3)
Dizziness (Vascular disorders) | 2 (2) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 5 (5) | 2 (2)
Heartburn (Gastrointestinal disorders) | 3 (3) | 7 (7) | 5 (5)
Low vitamin D (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 1 (1)
Nausea/vomiting (Gastrointestinal disorders) | 3 (3) | 7 (10) | 6 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No